CLINICAL TRIAL: NCT02177279
Title: Identification of Novel Bioactive Compounds in Wheat Bran
Brief Title: Bioactive Phytochemicals From Wheat Bran
Acronym: WB2001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Kellogg Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Wheat Bran 2001
Record Dates: First submitted 2014-06-19; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Bio-availability of Wheat Bran Phytochemicals in the Human Gut; Bio-availability of Wheat Bran Phytochemicals for the Systemic Circulation
Keywords: Wheat bran cereals, bran phytochemicals, phytochemicals bioavailability

ARMS (3):
- Visit A- 120g wheat bran cereals (Other): A morning vist where volunteers consumed 120g of wheat bran cereals with 125ml semi-skimmed milk
  Interventions: Other: Visit A high wheat bran
- Visit B-40g wheat bran cereals (Other): A morning vist where volunteers consumed 40g of wheat bran cereals with 375 ml semi-skimmed milk
  Interventions: Other: Visit B normal wheat bran
- Follow up-40g (8days), 120g (1day) wheat bran cereals (Other): Volunteers follow their normal diet but they were asked to consume 40g wheat bran cereals with 125 ml semi-skimmed milk for eight days and on day nine 120g wheat bran cereals with 375ml semi-skimmed milk
  Interventions: Other: Follow up normal (8days) and high (1day) bran consumption

INTERVENTIONS:
Other: Visit A high wheat bran
  Arms: Visit A- 120g wheat bran cereals
Other: Visit B normal wheat bran
  Arms: Visit B-40g wheat bran cereals
Other: Follow up normal (8days) and high (1day) bran consumption
  Arms: Follow up-40g (8days), 120g (1day) wheat bran cereals

SUMMARY:
There is a lot of evidence to suggest that eating a diet rich in cereals such as wheat bran are beneficial in protecting us from diseases such as heart disease, diabetes and cancer. It is still not clear exactly why this happens, but it is likely that the compounds which enter our bodies when we eat such products are responsible. In this study we plan to find out what these compounds are and where they are found. The investigators will do this by asking volunteers to eat a wheat-bran meal and then measuring the compounds that appear in blood, urine and stool samples over the next twenty-four hours. Once the investigators know how much and which compounds are present, we can then find out possible reasons why they are protective, for example by looking to see whether they are anti-inflammatory. We also plan to look at whether if having a diet which contains either a lot of wheat-bran products or very low amounts of these foods effects how they are absorbed by the body.

HYPOTHESIS: Wheat bran from ready-to-eat cereal has unique phytochemical profiles which are metabolized to compounds responsible for high cellular bioactivity imparting important health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be healthy males or females and aged between 18 and 55 years who have a documented low (less than 1 portion per week) or high (more than or equal 5 portions per week) consumption of wheat bran and are able to give informed consent.

Exclusion Criteria:

* are taking any medicines prescribed by their general practitioner
* are taking drugs to lower high cholesterol levels or high blood pressure
* regularly take analgesics, antipyretic or anti-inflammatories
* regularly take nutritional supplements
* have taken antibiotics in the last three months
* have given a large blood donation in last three months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Human bioavailability of benzoic acids and derivatives from wheat bran cereals | over 24 h
  The analysis of the benzoic acid and derivatives metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Human bioavailability of cinnamic acids and derivatives from wheat bran cereals | over 24h
  The analysis of the cinnamic acids and derivatives metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Human bioavailability of phenylpropanoid dimers from wheat bran cereals | over 24h
  The analysis of the phenylpropanoid dimers metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Human bioavailability of phenyl propionic acids from wheat bran cereals | over 24h
  The analysis of the phenyl propionic acids metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Bioavailability of benzaldehydes from wheat bran | over 24h
  The analysis of the benzaldehydes metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Human bioavailability of acetophenones from wheat bran cereals | over 24h
  The analysis of the acetophenones metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Human bioavailability of lignans from wheat bran cereals | over 24 h
  The analysis of the lignans metabolites in blood, urine, faecal samples after consumption of 40g and 120g wheat bran cereals, over 24 h period (change from baseline time 0h).
Short chain fatty acids profile after wheat bran consumption (acute) | 24 h
  Short chain fatty acids profile in faecal samples at 0h (baseline) and 24h after wheat bran consumption (40g and 120g).
Short chain fatty acids profile after wheat bran consumption (chronic) | 9 days
  Short chain fatty acids profile in in faecal samples at day 0 (baseline), day 5 (during 7 days consumption of 40g wheat bran cereals/day) and day 10 (after 120g wheat bran cereals consumption on day 9).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy R Russell, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen; Baukje de Roos, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen; Garry Duthie, Professor, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen; Jolene McMonagle, PhD, Principal Investigator — Kellogg Company; Reg Fletcher, PhD, Principal Investigator — Kellogg Company
Locations (1):
- Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Aberdeenshire, United Kingdom